CLINICAL TRIAL: NCT03966781
Title: A Randomized, Single-blinded, Single-center, Parallel-group, Sham-controlled, Prospective Trial of Combined Extracorporeal Shock Wave Lithotripsy and Endotherapy for Pain in Chronic Pancreatitis
Brief Title: Extracorporeal Shock Wave Lithotripsy and Endotherapy for Pain in Chronic Pancreatitis
Acronym: SCHOKE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Collaborators: Aalborg University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AIG/IEC28/04.2017-03
Record Dates: First submitted 2019-01-13; First posted 2019-05-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Chronic Pancreatitis; Chronic Pain
MeSH Terms: conditions — Pancreatitis, Chronic; Chronic Pain | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESWL followed by ERCP (Active Comparator): Patients enrolled in the active treatment group will be subjected to ESWL followed by ERCP and pancreatic duct stenting.
  Interventions: Procedure: ESWL; Procedure: ERCP
- Sham ESWL followed by sham ERCP (Sham Comparator): Patients enrolled in the sham treatment group will be subjected to sham ESWL followed by sham ERCP with no pancreatic duct intervention.
  Interventions: Procedure: Sham ESWL; Procedure: Sham ERCP

INTERVENTIONS:
Procedure: ESWL — ESWL will be conducted under epidural anesthesia. For epidural anesthesia, bupivacaine will be used to block the T6-T12 spinal segments. The patient's eyes will be lightly covered all along the procedure. Once epidural anesthesia is achieved, the patient will be given a light sedation and ESWL will be performed using a Dornier dual focus lithotripsy system providing a maximum of 5000 at the rate of 90 shocks per minute in over 1-2 days.
  Arms: ESWL followed by ERCP
Procedure: ERCP — Once ESWL is over, an endoscopic pancreatic sphincterotomy will be performed and complete stone removal will be attempted with subsequent stenting of the pancreatic duct in the presence of a pancreatic stricture (not detected on MRCP prior to enrolment) or in case of incomplete stone removal
  Arms: ESWL followed by ERCP
Procedure: Sham ESWL — In the sham/control group, patients will be given a transient superficial pin-prick sensation to give the feel of epidural anesthesia. After that the lithotripsy machine the will be switched on, without establishing any form of contact with the patients body.
  Arms: Sham ESWL followed by sham ERCP
Procedure: Sham ERCP — Following sham ESWL patientswill be subjected to sham ERCP to examine the papillary area, but no pancreatic ductal intervention will be performed.
  Arms: Sham ESWL followed by sham ERCP

SUMMARY:
Pain is a common symptom of chronic pancreatitis and remains a significant therapeutic challenge. In patients with pathological changes of the pancreatic duct, including stones and strictures, endoscopic procedures with or without preceding extracorporeal shock wave lithotripsy (ESWL) have been used with varying success to treat pain, but high quality evidence is lacking so support this practice. The main objective of this study is to investigate the pain-relieving effects of combined ESWL and endotherapy in patients with painful CP in comparison with sham treatment.

DETAILED DESCRIPTION:
Pain is the predominant symptom in patients with chronic pancreatitis (CP) and remains a considerable therapeutic challenge. In patients with pathological changes of the pancreatic duct, including stones and strictures, endoscopic procedures with or without preceding extracorporeal shock wave lithotripsy (ESWL) and surgery have been used with varying success to treat pain. The rationale for endoscopic therapy or surgical drainage procedures is based on the hypothesis that obstruction of the pancreatic duct leads to ductal hypertension and pain. However, clinical pain symptoms correlate poorly with pancreatic ductal morphology and the response to endoscopic or surgical treatment is unpredictable, with long term response rates ranging from 30-60%. The evidence for these treatments are, however, based on case-series and comparison between different procedures, while no prospective sham controlled trials have evaluated the effectiveness of invasive treatments for pain in CP. In addition, a marked placebo effect has been observed in most trials of painful CP and this, together with the natural history of disease, needs consideration when treatment effects are evaluated. Therefore, the rationale behind invasive treatments for pain in CP treatments can be questioned.

Recent meta-analyses have documented that the non-specific effects of surgery and other invasive procedures are generally large; particularly in the field of pain-related conditions. For example, arthroscopic meniscectomy for degenerative meniscal lesions has for many years been considered the state of the art treatment for this common condition. However, a high quality randomized controlled trial (RCT) and meta-analysis have not shown any differences in pain relieving effects between surgery and sham procedures for degenerative meniscal lesions. These findings challenge conventional wisdom and underline the necessity of properly conducted RCTs including a sham procedure, when the effectiveness of invasive procedures is evaluated.

Albeit endoscopic therapy or surgery are widely used for pain in CP these treatments are only effective in a subset of patients. An improved understanding of the mechanisms underlying pain in CP suggest that the pain etiology in most patients is multifactorial and, in addition to the proposed mechanical mechanisms for pain (ductal obstruction/hypertension), a large body of evidence support a ´neuropathic pain phenotype´ with abnormal processing in the peripheral and central neural pathways. This likely explains the variable response to endoscopic and surgical treatments and underline an unmet need for biomarkers to identify responders to the different treatment modalities.

Quantitative sensory testing (QST) can be used to investigate the state of the pain system; the technique is based on the rationale that different neural pathways and networks can be explored using standardized stimulation with simultaneous recording of the evoked pain response by psychophysical and/or objective methods. Due to spinal convergence between visceral afferents from the pancreas and somatic afferents from the Th10 skin dermatome, somatic QST can be reliable used to assess if the pain system is locally sensitized by nociceptive input from the pancreas (segmental sensitization). However, in many patients with chronic pain the pain system has become dysfunctional and has undergone a more universal sensitization. In such cases the QST profile of testing in several dermatomes together with specific test paradigms (temporal summation and assessment of descending inhibition) can be used to determine whether patients have abnormal central pain processing.

The hypothesis of the present study is that combined ESWL and endotherapy induce short term (3 months) and mid-term (6 months) pain relief in patients with CP compared to a sham procedure. In addition, the investigators hypothesize that QST can be used to predict the outcome of combined ESWL and endoscopic therapy. Hence, patients with evidence of abnormal pain processing are hypothesized to have a worse outcome to treatment compared to patients with segmental or no evidence of sensitization.

ELIGIBILITY:
Inclusion Criteria:

* Patients from the ages of 18 with a diagnosis of chronic calcific pancreatitis diagnosed using the Mayo Clinic diagnostic criteria. Both diabetic and non-diabetic patients will be allowed to enter the study.
* The patients must suffer from chronic abdominal pain characteristic for CP with a pain intensity >3 VAS on a 0-10 VAS and meet the criteria for chronic pain (pain ≥ 3 days per week in at least 3 months).
* Obstruction of the pancreatic duct due to intraductal stones with dilatation of the duct proximal to the obstruction, as determined by magnetic resonance cholangiopancreatography, abdominal computed tomography, or both.
* The patients must be able to read and understand the provided informed consent.
* Patients must personally sign and date informed consent document indicating that he/she has been informed of all pertinent aspects of the trial.
* Patients should be willing to comply with the scheduled visits, clinical and experimental assessment plan, and other trial procedures.

Exclusion Criteria:

* Patients with any clinically significant laboratory abnormalities that in the opinion of the investigator may increase the risk associated with trial participation or may interfere with the interpretation of the trial results.
* Previous history of pancreatic surgery, ESWL or ERCP.
* Patients with a pancreatic stricture on cross-sectional imaging prior to study enrolment
* Active alcohol or illegal drug dependencies.
* Patients with evidence or history of medical or surgical disease of importance for this study as judged by investigator.
* Patients must not suffer from painful conditions other than CP that make them unable to distinguish the pain associated with CP from chronic pain of other origin.
* Presence of pancreatic head mass, multiple strictures, large ascites, large fluid collections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
Change from baseline pain score at 3 months | 3 months after intervention
  The primary clinical endpoint is pain relief. Average and maximal daily clinical pain intensity scores will be recorded in a patient pain diary based on a 0-10 visual analogy scale (VAS), with registration of the baseline pain intensity scores the week prior to intervention and weekly recordings continued for a 3 months period after intervention. Mean values of pain scores will be calculated over 1 week to adjust for day-to-day variability in pain intensity. The difference in pain scores between patients receiving active treatment (ESWL and ERCP) and sham treatment are compared, with the primary comparison of average pain scores 3 months after intervention. Weekly telephone interviews from a study co-ordinator will be undertaken to facilitate accurate registration and compliance pain score).

SECONDARY OUTCOMES:
Ratio of responders versus non-responders | 3 and 6 months after intervention
  The ratio of responders versus non-responders defined by a decrease in the average clinical pain score (VAS) of 30% after 3 and 6 months compared to baseline.
Change in analgesic consumption | 3 and 6 months after intervention
  Change in analgesic consumption (if used) after 3 and 6 months compared to baseline
Hospitalization | 3 and 6 months after intervention
  Total number of hospitalizations during the study period after 3 and 6 months
Change in quality of life (EORTC-QLQ C 30) | 3 and 6 months after intervention
  Change in quality of life using the European Organization for Research and Treatment of Cancer Quality of Life questionnaire (EORTC-QLQ-C30) after 3 and 6 months compared to baseline
Changes in pain and physical functioning composite scores (BPI-sf) | 3 and 6 months after intervention
  Changes in pain and physical functioning composite scores of the modified brief pain inventory-short form (mBPI-sf) after 3 and 6 months compared to baseline
Patient Global Impression of Change | 3 and 6 months after intervention
  Patient Global Impression of Change (PGIC) after 3 and 6 months
Complications | 3 and 6 months after intervention
  Assessment of complications to interventions after 3 and 6 months
Change from baseline pain score at 6 months | 6 months after intervention
  This will be evaluated as described for the primary end-point
Pain free days after intervention | 3 and 6 months after intervention
  Difference in number of pain free days between groups after 3 and 6 months.
Change in anxiety and depression after intervention | 3 and 6 months after intervention
  • Difference in depression and anxiety scores of the Hospital Anxiety and Depression scale between groups after 3 and 6

OTHER OUTCOMES:
Quantitative sensory testing (characterization of pain processing) | 3 and 6 months after intervention
  The following experimental pain measures will be employed prior to intervention as well as 24-48 hours and 3 months after intervention to characterize changes in pain processing induced by the assigned procedures:
  * Muscle pressure stimulation (pancreatic viscerotome (Th10 ventral and dorsal) and control areas (C5, L1 and L4).
  * Bone pressure stimulation (tibia bone)
  * Temporal summation to repetitive pinprick stimulations of the pancreatic area (Th10) and control area (dominant forearm)).
  * Conditioned pain modulation (CPM).

CONTACTS AND LOCATIONS:
Locations (1):
- Asian Institute of Gastroenterology, Hyderabad, Andhra Pradesh, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Talukdar R, Olesen SS, Unnisa M, Bedarkar A, Sarkar S, Tandan M, Jagtap N, Darisetty S, Kiran S, Koppoju V, Lakhtakia S, Ramchandani M, Kalapala R, Gupta R, Singh VK, Rao GV, Reddy DN, Drewes AM. Extracorporeal Shock-Wave Lithotripsy and Endoscopy for the Treatment of Pain in Chronic Pancreatitis : A Sham-Controlled, Randomized Trial. Ann Intern Med. 2024 Jun;177(6):749-758. doi: 10.7326/M24-0210. Epub 2024 May 28. PMID 38801774
- [Derived] Olesen SS, Drewes AM, Gaud R, Tandan M, Lakhtakia S, Ramchandani M, Rao GV, Reddy DN, Talukdar R. Combined extracorporeal shock wave lithotripsy and endoscopic treatment for pain in chronic pancreatitis (SCHOKE trial): study protocol for a randomized, sham-controlled trial. Trials. 2020 Apr 16;21(1):338. doi: 10.1186/s13063-020-04296-0. PMID 32299454